# **Project Title**

Life story work for promoting relationship between older adults and live-in migrant caregivers: a randomized controlled feasibility trial.

This project was approved by the Research Ethics Committee of Tung Wah College on 24 Sep 2018.

Last updated: 13 Aug 2018

#### Abstract of research:

The relationship between older adults and live-in migrant caregivers is always challenged by weak emotional connectedness, ineffective communication, power struggling and unmet needs of both, that may lead to poor care quality and negatively influence their well-being. The aim of this study is to explore the feasibility to train live-in migrant caregivers to adopt Life Story Work for promoting the dyadic relationship with the older adults, through communication and negotiation, mutual understanding and expression of needs. This is a two-arm randomized controlled trial. The caregivers of the intervention group will receive training on life story work. Then they will be asked to create a life storybook of the older adult at home individually, with the support from the team. The caregivers in the control group will receive training on communication skills only, and will be asked to conduct social activities at home. Outcomes such as quality of relationship; well-being, depressive symptoms and level of loneliness of the older adults; and job satisfaction of the caregivers will be assessed at baseline, post-intervention and 3 months follow up. Focus group interviews will be conducted with the caregivers of the intervention group for soliciting their comments regarding to the intervention.

#### 1. The project aims and long-term significance:

(State the aims and identify the key issues and problems being addressed and the possible outcome of the research project, its relevance significance and value) (About 300 words)

There are approximately 21.5 million live-in migrant workers, and around 41% of them are employed in Asia (1). Among the 352 thousand live-in migrant workers in Hong Kong, at least 21% of them are caregivers of older adults (2). The 2016 Policy Address suggested a pilot scheme for training live-in migrant caregivers to take care of the older people in Hong Kong to meet the trend of Ageing in Place, and cope with the dreadful shortage of formal long-term care services (3). As such, Social Welfare Department of Hong Kong is now implementing an 18-month pilot scheme to train live-in migrant workers to care for older adults in order to improve the well-being of the older adults (4). However, there is no effective evidence-based intervention available for such caregiving arrangement, not only locally but also internationally. The common training for live-in migrant workers is about instrumental training, such as feeding and bathing (4). According to the Relationship-Centred Care Model, relationship is the core for good quality of care (5). Life story work have been tested effective in various settings for promoting the psychological well-being of older adults with/out dementia (6) (7), as well as proven useful in promoting mutual understanding and communication between caregivers and carerecipients (8).

## The project is of value in that:

- It is a pioneer study, which aims to promote relationship between live-in migrant caregivers and older adults to support good quality of care.
- The life story work is a skill that is easily learnt and adopted for promoting and sustaining good relationship that may impact on the well-being of caregivers and care-recipients.
- Reduce the needs of formal long-term care services by retaining the older adults to be cared at home.
- The life story work has a potential to be adopted by all types of caregivers (including formal and informal caregivers; live-in and live-out) for promoting the caregiver-care recipient dyadic relationship through communication and negotiation between the dyads, mutual understanding and expression of needs.

# 2. Objectives (State the objectives in point form):

- 1. Explore the feasibility to train live-in migrant caregivers to adopt life story work;
- 2. Explore the feasibility of trained live-in migrant caregivers to produce a life story book with the older adult at home; and
- 3. Provide preliminary evidence of efficacy of the life story work on improving dyadic relationship, psychosocial outcomes of the older adults, and satisfaction of caregivers.

# 3. Background of research and research plan and methodology: (Maximum 4 pages, excluding references)

[Summary of related work already done and outline of previous and alternative approaches to the problem

- (a) By others (give key references)
- (b) By the investigator(s) (give key references)
- (c) Progress report (for on-going projects)]

[Explain, in terms of the educated layman, the novel idea which you will be introducing to tackle the problem in question. Please include key references. Attach a draft questionnaire should the research plan involve a survey/interview.]

#### INTRODUCTION

Employing migrant workers as live-in caregivers for older adults is common around the world, particularly in the affluent countries (9). The relationship between the older adults and the live-in migrant caregivers (hereafter referred to as "caregivers") is unique and somehow ambivalent. Their relationship occasionally goes beyond the usual boundaries of formal employer-employee, but more companion-like or family-like (10) (11). In some studies, employers regarded the caregivers as "contractual or social" family members to describe the quasi-familial relationship (11) (12). This kind of relationship is always being challenged, especially coupled with the shared living arrangement as a risk factor for elder abuse (13). Both the older adults or caregivers are always portrayed themselves as victims or being maltreated (14). For example, the estimated prevalence rate of elder abuse is 15.7% globally (15), whereas that of Hong Kong was 21.4% (16). No family kinship relationship and past history together causes weak emotional connection (17). Because of the close living arrangement, caregivers are easily be asked to provide round-the-clock care that creates strain (18). More importantly, because of the language and cultural difference, and generation difference between the older adult and caregiver, creating difficulty in mutual understanding and effective communication (17) (19). Studies have consistently reported that older adults with cognitive impairment imposed even greater caregiving burden due to the disease related behavioural symptoms complicating the caregiving experience on the functional dependency (20) (21).

Poor caregiver-care recipient relationship have been shown causing poor care quality (5); poor well-being of both (22) (23); weak social support from the caregiver to the older adult who is already isolated because of frailty, leading to loneliness (24); and low satisfaction in caregivers (25). Hence, it is important to address this unique caregiver-care recipient relationship, of which is theoretically interdependent, and is central to the caregiving process. Donabedian suggested that good care is dependent not only on technical care, but also on a good interpersonal processes, which is a shared endeavor (26).

Relationship-centred care is an emergent concept that goes beyond the individualized task-centred and person-centred models by acknowledging the personhood in the caring process (i.e. not only the care recipient) (5). It emphasizes the reflection of the needs of caregivers alongside the needs of the older adult, in order to create a more participatory approach to achieve better care outcomes (5). In a relationship-centred care approach, it encompasses at least four important elements: anticipating needs of older adults and caregivers; negotiation between the dyad; shared understandings; and recognizing the contribution. By applying the relationship-centred care approach, older adults would satisfy with the care they receive. Studies suggested caregiver to adopt a life story approach to relate with older adult; and to get to know his/her and to ensure 'what matters' to the older adult is captured and transferred into everyday care (5) (27) (28).

Life story work (LSW) gives people an opportunity to share their memories and talk about their life experience (29). LSW highlights a person's unique life history and provides a greater insight into a person's needs and behaviours (30). Stories are threads that weave together the life of an older adult, and are the raw material from which the sense of self emerges (31). Thereby, connecting the past and present life events allows older people to preserve their own identity and affirming a sense of agency (32). People with dementia (PWD) are at higher risk of losing their identity because of the fractured connections between life events. LSW is therefore

a traditional approach to re-establish the positive self-identity for PWD from mid to later stages, albeit without much details about its effect for PWD in early stage (32). The preferred format of LSW is a life story book (LSB) (32). Attentive listening through LSB creation permits caregivers access to understand the older adults' meanings, beliefs, and values that enriches relationships (33). Expressions of concern and sage comments restore a reciprocity of caring (33). Creating the LSB together also allows the recognition of commonalities and differences and begins a transformation in the process of how the caregiver and older adult come to know and connect with one another (33).

Studies have shown that creation of LSB can improve psychosocial outcomes, such as well-being, depressive symptoms, and loneliness by valuing one's life and feeling of connectedness (7) (34). Literature also provides strong evidence showing that the creation of LSB can promote understanding of the older adults and improve communication between caregiver and older adults when adopted in nursing homes (27) (28) (35) (36). Applying the relationship-centred care model, LSB can be viewed as an intervention for promoting care quality, through communication and negotiation between the dyads, mutual understanding, and expression of needs (5). Therefore, we are proposing to train live-in migrant workers to adopt LSW to improve their relationship with the older adults.

## **METHODS**

The aim of this study is to explore the feasibility to train live-in migrant caregivers to adopt life story approach and how the trained live-in migrant caregivers produce the life storybook with the older adults; and provide preliminary evidence of efficacy of the intervention on promoting relationship, psychosocial outcomes of the older adults and caregivers, and caregiver satisfaction.

**Design:** Two-arm single-blinded randomized controlled feasibility trial. The outcomes will be measured at baseline (T0), immediately post-intervention (T1), and 3-month follow up (T2). To review the acceptability and the practical concerns of training caregivers to adopt life story approach for promoting the relationship with older adults, all caregivers in the intervention group will be invited to participate focus-group interview at T1. Recruitment, retention, safety issues will be monitored.

Setting and participants: St James Settlement (SJS) District Elderly Community Centre, Wan Chai district is the collaborator of this project, of which has a long experience to work with caregivers and older people (see appendix I for the collaboration agreement). The dyads of older adult and the caregiver will be the target population. The older adults should be aged 60 or above; community-dwelling; and being cared by the participating caregivers. Those who is unwilling to create the LSB with the caregivers; not verbally communicable; and diagnosed with serious psychiatric illness or terminal illnesses will be excluded. The caregivers should have been working for the older adults for more than 6 months, so that basic trust is established. In order to ensure the caregivers are competent to follow the protocol of LSB creation, he/she should have at least completed primary education and be communicable in either English or Cantonese. The training will be taken place in Tung Wah College or venues provided by SJS and the creation of the LSB will be done at the participant's home.

Sample size: As this is not a hypothesis testing trial, a formal power analysis is not required. However, a minimum of 10-20 dyads per group will be enough for meaningful group comparison (37). We aim to recruit 50 dyads in total in this study, given that we anticipate less than 20% of drop-out, and have a minimum of 20 dyads per arm. For the focus group interview, all the participated caregivers in intervention group will be invited to form four focus groups.

Recruitment: Convenience sampling will be employed. St James Settlement (SJS) will refer potential caregiver participants, and will assist to invite the older adults cared by the potential caregiver participants in this project. Information sheet about the study will be given to the participating dyads. We anticipate the recruitment process will take around 6 months to reach the target sample size.

*Intervention:* The goal of the intervention is to promote the relationship between the older adults and caregivers through the creation of LSB, in which allows communication and negotiation between the dyads, mutual understanding, and expression of needs. The caregivers of the intervention group will receive training (four weekly 3-hour session) about life story approach by a part-time registered social worker with at least three years of working experience working with older people and have basic knowledge about the LSW (refer

to appendix II for the caregiver training protocol). After training, they will be asked to produce the LSB individually at home with the older adults, with the assistance of a trained student assistant / research assistant (RA) served as an interpreter. The protocol of LSB creation is validated in Hong Kong by Prof. Claudia Lai (38) (refer to appendix III for the intervention protocol and appendix IV for the training protocol on student helpers and RA). Four to six 60-minute scheduled sessions will be needed for the older adult and the live-in migrant care worker to discuss and produce the LSB at home. The LSB would contain two elements: (1) the development of the older adults over the course of his/her lifetime (i.e. from childhood to old age); and (2) the psychosocial development and ways of life of the older adults (e.g. education, marriage, career, and hobbies). The product of the intervention will be a written story with pictures or other memorabilia that are meaningful to the older adults. There is no limitation on the number of words, pages, and pictures.

Control condition: The caregivers who have randomly assigned into the control group will receive communication skills training (two 3-hour sessions) offered by another registered social worker with at least three years of working experience working with older people. They would not receive any additional training on LSW. However, to control the possible social interaction effects on the dyadic relationship and wellbeing, the caregivers of the control group will be asked to conduct a self-selected social activity with the older adult at home individually for four times weekly with the assistance of a student assistant served as an interpreter. The social activity can be chess playing, art making or game playing.

**Measures:** A trained research assistant will be responsible to collect demographic data and assessing the outcomes at T0, T1 and T2. The P.I. will conduct the focus group interviews with the caregiver participants as soon as the intervention is completed. Outcomes measuring tools and interview questions are listed in appendix V.

Primary outcomes: Quality of the caregiver-care recipient relationship

As the relationship between the dyads can be viewed differently from two individuals, both participants will be asked to answer the questions related to the relationship quality. It will be measured with the 4-item Lawrence Quality of the caregiver-care recipient relationship scale (39), and another 4-item scale developed by a study evaluating the relationship quality of live-in migrant caregivers with older adults (17). General closeness, communication, similarity of views about life, and degree of getting along will be captured by the first scale, while the feeling of closeness, getting along well, understanding each other, and an overall rating of the quality of the relationship will be reflected by the latter scale.

Secondary outcomes:

Loneliness of the older adult: Chinese version of 6-item De Jong Gierveld Loneliness Scale (40)

Depressive symptoms of the older adult: Chinese version of 15-item Geriatric Depression Scale (41)

Well-being of the dyad: General Health Questionnaires 12-item (42)

Satisfaction of caregiver: Care Work Satisfaction Scale (43)

Possible confounders: Dependency level of older adult: Modified Barthel Index (44)

Feasibility indicators: Ease of recruitment, adherence rate, drop-out rate, satisfaction of the dyads on the intervention will be assessed.

Qualitative process evaluation: The focus group interviews will be conducted for describing the caregiver's learning process and their interactions with older people on the creation of LSB. Upon informed consent from the participants, the interviews will be audio recorded and transcribed verbatim. The facilitator will encourage participant caregivers to interact in order to uncover various aspects in learning and implementing LSB. The following prompting questions will be asked in the focus group interviews with the caregivers by narrowing down from general questions to focus questions (45):

- 1. Would you please tell me your experiences/opinions with regard to learning and participating in the intervention?
- 2. Would you please tell whether participating in the intervention has made a difference or not in relation to your relationship with the live-in migrant care worker/older adult?
- 3. What were the challenges in conducting LSB with older adults?
- 4. How does the employer-employee relationship affect your communication and production of LSB with older adults? Probing: Or is it a concern for you?

5. Any other comments/suggestions based on your participation in the intervention? *Fidelity monitoring:* 

A checklist has been developed for monitoring the compliance of the participants during the intervention (See Appendix VI).

**Randomization**: After obtaining the written informed consent from both the older adult and caregivers, each dyad will be asked to toss a coin for group assignment.

Data analyses: SPSS version 24 for Windows will be used for all statistical analyses. All the statistical analysis will be based on intention-to-treat principles. To examine group differences at baseline, independent t-test and Mann-Whitney U test will be performed with all continuous demographic and outcome variables if they are normally or non-normally distributed respectively. Chi square test will be done for comparing categorical variables. To examine group differences at post (T1) and follow up (T2) assessment, individual analyses of covariance (ANCOVAs) will be performed with baseline treatment outcome scores used as the covariate. Effect sizes will be calculated using Cohen's d for each outcome measure. The focus group interview will be transcribed verbatim for content analysis (46). The analysis will focus on identifying and describing the facilitators and barriers for participants to learn the creation of LSB and their perceived challenges and perceived benefits in implementing LSB with older adults. Transcription will be open coded. Codes with similar meanings will be translated into categories. Codes and categories will be compared and contrast between focus groups in order to identify the patterns in the learning process of LSW and implementation of LSB. These patterns will be represented by themes of higher level of abstraction.

*Safety and monitoring:* The trial will be overseen by the project team and the staff of the SJS. The team will be responsible for monitoring the progress of the study and the safety issues. All adverse event will be recorded and reported to the College and the SJS.

Ethical consideration: Ethical approval will be obtained from the College and the SJS. Participation in the study will be entirely voluntary. Informed written consent will be sought from both the older adult and caregiver participants. The caregivers will be asked to sign a confidentiality agreement that the information collected during the LSB creation will be kept confidential. When the older adults encounter any emotional disturbance during the production of the LSB, the team will follow up with the issues and make necessary referrals.

#### TIMELINE

| | _ | | | | | | | | Mar-19 | Apr-19 | | | | | | _ | | | | | | _ | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Month | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | B | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| | Preparation & Orientation | | | | | | | | | | | | | | | | | | | | | | | | |
| Orientation and training to | | | | | | | | | | | | | | | | | | | | | | | | | |
| research personnel Meetings with study sites | | | _ | | | | | | | | | | | | | | | | | | | | | | - |
| to finalize logistics | | | | | | | | | | | | | | | | | | | | | | | | | |
| Dinama: rogsaco | | | | | | | | | | _ | nrolme | | | | | | | | | | | | | | |
| District of the second | | | | | | | | | | - | iii olme | III. | | | | | | | | | | | | | |
| Bigibility screening | | | | | | | | | $\vdash$ | | | | | | | | | | | | | | | | <u> </u> |
| informed consent | | | | | | | | | | | | | | | | | | | | | | | | | |
| Group allocation | | | | | | | | | | | | | | | | | | | | | | | | | |
| | | | | | | | | | | Int | terventi | ons | | | | | | | | | | | | | |
| Intervention group | | | | | | | | | | | | | | | | | | | | | | | | | |
| receiving standard training | : | | | | | | | | | | | | | | | | | | | | | | | | |
| +life story approach | | | | | | | | | | | | | | | | | | | | | | | | | |
| Control group receiving | | | | | | | | | | | | | | | | | | | | | | | | | |
| standard training | | | | | | | | | | | | | | | | | | | | | | | | | <u> </u> |
| Intervention group producing ISB at home | | | | | | | | | | | | | | | | | | | | | | | | | |
| individually<br>producing constraine | | | | | | | | | | | | | | | | | | | | | | | | | |
| Control group conducting | | | | | | | | | | | | | | | | | | | | | | | | | |
| social activities at home | | | | | | | | | | | | | | | | | | | | | | | | | |
| individually | | | | | | | | | | | | | | | | | | | | | | | | | |
| - | | | | | | | | | | As | sessme | nts | | | | | | | | | | | | | |
| TD Assessment | | | | | | | | | | | | | | | | | | | | | | | | | |
| T1 Assessment | | | | | | | | | | | | | | | | | | | | | | | | | |
| TZ Assessment | | | | | | | | | | | | | | | | | | | | | | | | | |
| | | | | | | | | | | Proje | ct Comp | letion | | | | | | | | | | | | | |
| Data cleaning and analysis | | Π | | Π | | | | | | rioje | CC COMP | HELIOII | | | | | | | | | | | | | |
| Report and manuscript | | | | | | | | | $\vdash$ | | | | | | | | | | | | $\vdash$ | | | | <del></del> |
| writing | | | | | | | | | | | | | | | | | | | | | | | | | |
| | | | | | | | | | | | | | | | | | | | | | | | | | <u> </u> |

P.I. has extensive research work with the live-in migrant caregivers caring older adults. He has identified the needs of supportive intervention these caregivers in his research, in order to promote the unique relationship with the older adults. Co-I Dr Cheung has conducted several projects adopting dyadic interventions such as music intervention (47) (48)and play intervention (49) for older adults with dementia and their caregivers. She has strong competency in conducting RCT on dyadic intervention.

## **ANTICIPATING PROBLEM**

We are confident that we can recruit participants to the target number. However, if SJS cannot recruit enough caregivers to this project, other NGOs working with migrant workers and older people will be invited to participate in this project. The Co-Is (Dr. Cheung & Prof. Fung) have solid research collaborating relationship with the other organizations working with older people while the P.I. has solid relationship with organizations working with migrant workers.

#### References

- 1. **International Labour Organization.** Working conditions and attitudes experienced by migrant domestic workers in Thailand and Malaysia. Thailand: International Labour Organization, 2016.
- 2. **Legistlative Council Commission.** Foreign domesitc helpers and evolving care duties in Hong Kong. Hong Kong: Legislative Council Commission, 2017.
- 3. **The HKSAR Government.** 2016 Policy Address. [Online] 2016. [Cited: June 15, 2018.] https://www.policyaddress.gov.hk/2016/eng/.
- 4. **Social Welfare Department, HKSAR.** *Social Welfare Department.* [Online] 2018. [Cited: June 15, 2018.] https://www.swd.gov.hk/en/index/site\_pubsvc/page\_elderly/sub\_psfdh/.
- 5. Wilson, C.B. Caring for older people: A shared approach. London: SAGE Publications, 2013.
- 6. The functions and value of reminiscence for older adults in long-term residential care facilities. **Henkel, L.A., Kris, A., Birney, S., Krauss, K.** 3, 2017, Memory, Vol. 25, pp. 425-435.
- 7. Does life story work improve psychosocial well-being for older adults in the community? A quasi-experimental study. Lai, C.K.Y., Igarashi, A., Yu, C.T.K., Chin, K.C.W. 1, May 2018, BMC Geriatrics, Vol. 18.
- 8. Life story work in health and social care: systematic literature review. McKeown, J., Clarke, A., Repper, J. 2, July 2006, Journal of Advanced Nursing, Vol. 55, pp. 237-247.
- 9. The perspective of employers/families and care recipients of migrant live-in caregivers: a scoping review. Salami, B., Duggleby, W., Rajani, F. 6, November 2017, Health and Social Care in the Community, Vol. 25, pp. 1667-1678.
- 10. When foreign domestic helpers care for and about older people in their homes: I am a maid or a friend. **Ho K.H.M., Chiang, V.C.L., Leung, D., Ku, B.H.B.** January 2018, Global Qualitative Nursing Research, Vol. 5, pp. 1-10.
- 11. Live-in foreign domestic workers and their impact on Hong Kong's middle class families. Chan, A.H.N.
- 4, December 2005, Journal of Family and Economic Issues, Vol. 26, pp. 509-528.
- 12. Negotiating the social family: migrant live-in elder care workers in Taiwan. Lin, S., Bélanger, D. 3, 2012, Asian Journal of Social Science, Vol. 40, pp. 295-320.
- 13. **World Health Organization.** Elder abuse. *World Health Organization*. [Online] 2018. [Cited: June 20, 2018.] http://www.who.int/news-room/fact-sheets/detail/elder-abuse.
- 14. Abuse is in the eyes of the beholder: using multiple perspectives to evaluate elder mistreatment under round-the-clock foreign home carers in Israel. **Ayalon, L.** 3, April 2011, Ageing & Society, Vol. 31, pp. 499-520.
- 15. Elder abuse prevalence in community settings: A systematic review and meta-analysis. Yon, Y, et al. 2, 2017, The Lancet, Vol. 5, pp. e147-e156.
- 16. Prevalence and correlates of intimate partner violence among older Chinese couples in Hong Kong. Yan, E and Chan, K L. 2012, Int Psychogeriatr, Vol. 24, pp. 1437-46.
- 17. Like one of the family? Understanding relationships between migrant live-in care workers and older care recipients in Israel. **Teshuva**, **K.**, **Cohen-Mansfield**, **J.**, **Iecovich**, **E.**, **Golander**, **H.** February 2018, Ageing & Society, Vol. Ahead of print, pp. 1-22.
- 18. *A job with no boundaries. Home eldercare work in Italy.* **Degiuli, F.** 3, August 2007, European Journal of Women's Studies, Vol. 14, pp. 193-207.

- 19. Understanding and managing intergenerational conflict: An examination of influences and strategies. Urick, M.J., Hollensbe, E.C., Masterson, S.S., Lyons, S.T. 2, April 2017, Work, Aging and Retirement, Vol. 3, pp. 166-185.
- 20. Multivariate models of subjective caregiver burden in dementia: A systematic review. van der Lee, J., Bakker, T.J.E.M., Duivenvoorden, H.J., Droes, R. May 2014, Ageing Research Reviews, Vol. 15, pp. 76-93.
- 21. Caregiver burden for informal caregivers of patients with dementia: A systematic review. Chaio, C.Y., Wu, H.S., Hsiao, C.Y. 3, September 2015, International Nursing Review, Vol. 62, pp. 340-350.
- 22. Caregivers' relationship closeness with the person with dementia predicts both positive and negative outcomes for caregivers' physical health and psychological well-being. Fauth, E., Hess, K., Piercy, K., Norton, M., Corcoran, C., Rabins, P., Lyketsos, C., Tschanz, J. 6, May 2012, Aging & Mental Health, Vol. 16, pp. 699-711.
- 23. Interpersonal effects of suffering in older adult caregiving relationships. Monin, J.K., Schulz, R. 3, 2009, Psychology and Aging, Vol. 24, pp. 681-695.
- 24. Correlates of social and emotional loneliness in older people: evidence from an English community study. **Dahlberg, L., McKee, K. J.** 4, May 2014, Aging & Mental Health, Vol. 18, pp. 504-514.
- 25. Determinants of job satisfaction in foreign domestic helpers caring for people with dementia in Hong Kong. Bai, X., et al. 5, 2013, Health and Social Care in the Community, Vol. 21, pp. 472-479.
- 26. The quality of care. How can it be assessed? Donabedian, A. 12, 1988, JAMA, Vol. 260, p. 1743.
- 27. Using biography to enhance the nursing care of older people. Clarke, A. 7, April 2000, British Journal of Nursing, Vol. 9, pp. 429-433.
- 28. Life stories and biography: a means of connecting family and staff to people with dementia. **Kellett, U., Moyle, W., McAllister, M., King, C., Gallagher, F.** 11-12, June 2010, Journal of Clinical Nursing, Vol. 19, pp. 1707-1715.
- 29. Life story work in health and social care: systematic literature review. McKeown, J., Clarke, A., & Repper, J. 2, July 2006, Journal of Advanced Nursing, Vol. 55, pp. 237-247.
- 30. Valuing the person's story: use of life story books in a continuing care setting. Wills, T., Day M.R. 3, 2008, Clinical Interventions in Aging, Vol. 3, pp. 547-552.
- 31. Explorations of narrative identity. **Polkinghorne, D.E.** 4, 1996, Psychological Inquiry, Vol. 7, pp. 363-367.
- 32. *Life story resources in dementia care: A review.* **Kindell, J, et al.** 3, 2014, Quality in Ageing and Older Adults, Vol. 15, pp. 151-161.
- 33. Story sharing. restoring the reciprocity of caring in long-term care. Heliker, D. 7, July 2007, Journal of Psychosocial Nursing, Vol. 45, pp. 20-23.
- 34. The effects of reminiscence therapy on psychological well-being, depression, and loneliness among the institutionalized aged. Chiang, K. J., Chu, H., Chang, H. J., Chung, M. H., Chen, C. H., Chiou, H. Y., Chou, K. R. 4, April 2010, International Journal of Geriatric Psychiatry, Vol. 25, pp. 380-388.
- 35. Life story work sees the person beyond the dementia: A project to evaluate life story work, and how it helped care professionals and family carers as well as people with dementia. **Batson, P., Thorne, K., Peak, J.** 3, 2002, Dementia, Vol. 10, pp. 15-17.

- 36. Seeing the person behind the patient: enhancing the care of older people using a biographical approach. Clarke, A., Jane Hanson, E., & Ross, H. 5, September 2003, Journal of Clinical Nursing, Vol. 12, pp. 697-706.
- 37. Considerations in determining sample size for pilot studies. **Hertzog, M.A.** 2, 2008, Research in Nursing \* Health, Vol. 31, pp. 180-191.
- 38. Lai, C.K.Y. *Improving the quality of life for nursing home residents with dementia: a life story approach.* s.l.: Unpublished dissertation. TheUniversity of Hong Kong., 2004.
- 39. Quality of the caregiver—care recipient relationship: Does it offset negative consequences of caregiving for family caregivers? Lawrence, R. H., Tennstedt, S. L., Assmann, S. F. 1, March 1998, Psychology and Aging, Vol. 13, p. 150.
- 40. Validation of the Chinese translation of the 6-item De Jong Gierveld Loneliness Scale in elderly Chinese. Leung, G. T. Y., de Jong Gierveld, J., & Lam, L. C. W. 6, December 2008, International Psychogeriatrics, Vol. 20, pp. 1262-1272.
- 41. Chi, I., Yip, P. S., Chiu, H. F., Chou, K. L., Chan, K. S., Kwan, C. W., ... & Caine, E. (2005). Prevalence of depression and its correlates in Hong Kong's Chinese older adults. Chi, I., Yip, P.S., Chiu, H.F., Chou, K.L., Chan, K.S., Kwan, C.W., Conwell, Y. and Caine, E. 5, May 2005, Ther American Journal of Geriatric Psychiatry, Vol. 13, pp. 409-416.
- 42. **Golderberg, D. Williams, P.** A user's guide to the General Health Questionnaire. Windsor, UK: NFER-Nelson, 1988.
- 43. *Measuring the impact of informal caring*. **Orbell, S., Hopkins, N., Gillies, B.** 2, June 1993, Journal of Community & Applied Social Psychology, Vol. 3, pp. 149-163.
- 44. *Improving the sensitivity of the Barthel Index for stroke rehabilitation*. **Shah, S., Vanclay, F., Cooper, B.** 8, January 1989, Journal of Clinical Epidemiology, Vol. 42, pp. 703-709.
- 45. **Kruger, R A and Casey, M A.** Focus group interviewing. [ed.] K E Newcomer, H P Hatry and J S Wholey. *Handbook of Practical Program Evaluation*. 4th. Hoboken, NJ: Jossey-Bass, 2015, pp. 506-534.
- 46. *The qualitative content analysis process.* **Elo, S and Kyngäs, H.** 1, 2008, Journal of Advanced Nursing, Vol. 62, pp. 107-115.
- 47. Translational research on a dyadic approach to the music-with-movement intervention for people with dementia and their families. Lai, C.K.Y., Lai, D.L.L., Cheung, D.S.K., Chan, L.C.K. 7, July 2017, Alzheimer's & Dementia: the Journal of the Alzheimer's Association, Vol. 13, p. 1469.
- 48. Interdisciplinary collaboration in the use of a music-with-movement intervention to promote the wellbeing of people with dementia and their families: Development of an evidence-based intervention protocol. Lai, C.K.Y., Lai, D.L.L., Ho, J.S., Wong, K.K.Y., Cheung, D.S.K. 1, March 2016, Nursing & Health Sciences, Vol. 18, pp. 79-84.
- 49. Play Intervention for Dementia for promoting cognitive functions: a feasibility study. Cheung, DSK, Li, BY, Lai D, Yu, C.T.K., Leung, A, Tsang KT. 2018, Under review.

#### **Research Project Cooperation Agreement**

If Dr. Ken Ho, Assistant Professor of the School of Nursing at Tung Wah College, successfully applies for funding from the College Research Grant and conducts a research project (Life story work for promoting relationship between older adults and live-in migrant caregivers: a randomized controlled feasibility trial), the organization is willing to become a partner and provide the following assistance:

- Assist in the referral of Foreign Domestic Helpers and older adults to the research team;
- · Assist in the provision of space for conducting training;
- Assist in the promotion of the research project to other related community service providers.

| (Stamp) |
|------------------------------------------------|
| 聖雅各福群會<br>灣仔長者地區中心<br>Strict Elderly Community |

\*Name of Organization:

Date: 36/6/2018-

| S7. JA | MES' SETTLE | EMENT 1 | WAN | CHAI | DECC |
|-----------|-------------|---------|-----|------|------|
| n-charge: | NANG: | Pul ju | NG | | |
| Position: | SENIOR | MANAGE | R | | |

#### Training protocol for live-in migrant caregivers of older adults

Modified from Lai, C.K.Y. (2003). Improving the quality of life for nursing home residents with dementia: a life story approach. Dissertation: The University of Hong Kong.

#### Contents

- a. Basic knowledge and techniques required for leading LSB group
- b. Activity guidelines
- c. How to handle activity-related problems
- d. How to gain support from the family members of older adults

#### Basic knowledge and techniques required for leading LSB group

The live-in migrant caregivers are living together with the older adult for at least 6 months. They are expected to be proficient in the following basic skills:

- 1. Basic communication skills
- 2. Skills for communicating with their older care-recipient
- 3. Basic skills for communicating with older adult with mild dementia (if their older care-recipients are person with mild dementia)
- 4. Basic skills for managing the emotional and behavioural problems of the older care-recipient with/out dementia

#### **Activity guidelines**

The following are guidelines required specially for the purpose of this study.

#### Session 1:

- 1. Recognize the best way of addressing him/her.
- 2. Explain the objectives, contents usage, period and times of the activity.
- 3. Establish rapport to explain the roles of each party, emphasize that the LSB is produced by co-operation and the importance of his/her commitment. For example, the older adult may provide personal information or photos, choose or affix pictures, etc., whereas the caregiver may collect pictures and type captions.
- 4. Ask the older adult if there are any doubts about or problems with the activity.
- 5. Invite the older adult to choose a photo album from different colors.
- 6. Collect information about the older adult.
- 7. Conclude and show appreciation for the performance of the older adult.
- 8. Discuss and confirm the date and time for the next meeting.

#### Session 2-5:

1. Briefly introduce the activity. (As a revision, because the older adult may forget)

- 2. Put the collected photos, pictures and typed words according to the information provided by the older people into the photo album. Let the older adult read it and invite him/her to choose the right photos/pictures to put into the LSB.
- 3. Collect other information about the older adult.
- 4. Conclude and show appreciation for the older adult's performance.
- 5. Discuss and confirm the date and time for the next meeting.
- 6. In session 5, please remind the older adult that the next meeting will be the last session.

#### Session 6 (last session):

- 1. Briefly introduce the activity and remind the older adult that this is the last session of the activity. (As a revision, because the older adult may forget)
- 2. Put the collected photos, pictures and typed words and documents according to the information provided by the older people into the photo album. Let the older adult read it and invite him/her to choose the right photos/pictures or typed words to put into the LSB.
- 3. Review the whole LSB with the older adult.
- 4. Discuss how to use the LSB.
- 5. Conclude, show appreciation for the older adult's performance, and thank him/her for participating.
- 6. According to the arrangement made previously, hand the LSB to the older adult for storage.
- 7. Inform family members if necessary, to notify them of the completion of the LSB.

#### Points to Note:

- 1. Understand the problems and needs of the older adult and give appropriate guidance or assistance, e.g. if the older adult has a hearing impairment, then a hearing aid should be used.
- 2. Take account of the abilities of the older adults in choosing the style of words, pictures and photos, as well as adjusting his/her participation level and the concentration on what he/she can and cannot do, e.g. cutting and pasting, deciding where and how to affix the pictures and what other contents should be put into the LSB.
- 3. The most important is allowing the older adult to produce his/her LSB with you, instead of you making it for the older adult on your own.
- 4. Pay attention to the older adult's performance, interests and feelings, give him/her more consolation and encouragement as appropriate, and process the shared contents with flexibility.
- 5. Encourage the older adult to participate actively and show appreciation to him/her instantly.
- 6. Concentrate on discussing the positive experiences.
- 7. The caregiver's performance will also affect the older adult, therefore it can influence and encourage the older adults to join in if the caregiver can show participation, enthusiasm, or share his/her experiences appropriately.
- 8. Enquire as to how the LSB will be stored by the older adult.

Guideline to follow when the older adult speaks of unpleasant experiences in the past and becomes sad

- 1. There may be occasions on which, when discussing events in the past, the recall of unpleasant events by the older adults may bring back strong emotions. Therefore, the caregivers should always be sensitive to the expression and needs of the older adults.
- 2. Preparation beforehand is useful but may not always cover all sensitive areas that the older adult may react to.
- 3. When the older adult shows any signs of reluctance in talking about certain categories in the LSB protocol, the caregiver should be mindful of how to approach the topic. If it is a sign of sadness and the older adult is keen to discuss the topic further, it is only ethical for the discussion to continue.
- 4. It is also possible for the caregiver to divert attention from this topic if the older adult shows strong feelings about topic. After the session, it is then possible to collect some background information from the family, to gain some insights as to the nature of the problem and whether it is appropriate for the sessions to continue.
- 5. If it is a hurtful, traumatic experience that is being recalled, then it should not be included in the LSB. The production of the LSB is supposed to be an enjoyable event. It is neither an integrated life review, nor a therapy for resolution of previous conflicts. It is a structured recollection of a person's life history and, through the processes of producing it, an activity that provides opportunities for communication and interaction, and to help the caregiver to get to know the older adult better.
- 6. Should the older adult show signs of not letting go of the topic and of being upset for more than a brief while, s/he needs further support. The family members need to be informed and should maintain continual assessment. Seeking help from the research team for counseling and emotional support to older adult is appropriate when needed.

#### How to gain family members' support and co-operation

- 1. Introduce the life story book activity and explain the usefulness of the information provided by him/her.
- 2. Enquire whether the family member can provide some photos of the resident to affix into LSB; however, remind the family members that the photos provided should not be irreplaceable.
- 3. Show appreciation to the help of family members.

#### **Life Storybook Intervention Protocol**

Modified from Lai, C.K.Y. (2003). Improving the quality of life for nursing home residents with dementia: a life story approach. Dissertation: The University of Hong Kong.

#### 1. What is a life story?

A biography or life story in general refers to the history of an individual, a record of his/her life.

#### 2. How is a life story defined in this study for participants?

The term life story was defined in a generic and global sense, referring to glimpses of an individual's life, including reminiscence, rather than to a biography or an entire life story.

#### 3. Possible uses of an life storybook (LSB):

- a. An opportunity for the older adult to share with live-in migrant caregiver
- b. To encourage the older adult to interact with live-in migrant caregiver
- c. As reference for care planning for the older adult
- d. To provide emotional support and a sense of security through introducing a positive social environment for interaction
- e. Through reminiscing, to re-validate the worth of self as an unique individual
- f. To enhance self-esteem by re-discovering achievements in the past

#### 4. Book format

- a. Can be produced in many different styles and formats. LSBs appear to be the most meaningful when they are written in the first person.
- b. Drawings, maps, clippings, brochures, or anything creative that can be affixed to the album can be used.
- c. The older adults should not be giving up any treasured pictures or memorabilia. These items can be scanned or photographed.

#### 5. Contents suggestions

- a. Attention must be paid to what seems to interest the older adult. The best topics are the ones to which the older adult shows the most positive response. Input from family and friends is also important, as they know the older adult best.
- b. Although a standardized approach is adopted, the book can start or stop during any period of the older adult's life history. The choice may be dependent upon the older adult.
- c. The following suggested outline is by no means exhaustive. For the prompting questions under each category, please refer to Table 1.
  - · Family, roots/ancestry

- Religion
- Childhood
- Education
- Marriage
- Places lived
- Close friends/neighbors
- Work history
- Military history
- · Awards received
- Lifestyle
  - Interest and hobbies
  - Travel
  - Favorite foods, recipes
  - Holidays/festivals/seasons of the year
  - Involvement in clubs and groups, positions of leadership
  - Volunteer experiences or service organizations
  - Politics
  - Interest in literature and reading
  - Interest in music and creative arts
  - Animals and pets
- 6. Key points when working on the LSB with the older adult
  - a. Always be curious about the life story of the older adult so that s/he will be more willing to share.
  - b. Pictures and painting can also be used to help the older adult to recall memories
  - c. Be patient and allow ample time for older adults to respond
  - d. Offer plenty of opportunities for older adults to comment on the book in the process of production; provide lots of opportunity for involvement in the production processes, such as choosing pictures, cutting newspapers, and sticking the items onto the album.
  - e. Provide positive feedback as needed.
  - f. Be sensitive to the likes and dislikes, changing moods, needs and capabilities of the older adult, and be flexible. It is not appropriate to make the older adult, and be flexible. It is not appropriate to make the older adult perform any task or complete the session if s/he is unwilling.
  - g. It is fine for the live-in migrant caregiver to share their life story with the older adult that enhance mutual communication.
- 7. Guidelines for use of the produced LSB

- a. In general, the goal for the live-in migrant caregivers is increased sensitivity and understanding as they learn about the older adult's life history and the ability to apply the information to the current caregiving experience.
- Encourage the older adult to read phrases and captions under each picture or item in the LSB.
   Phrases or captions are useful because they can also be read by other relatives if need, as these are self-explanatory for those who may be reading the LSB for the first time, such as their grandchildren.
- c. Enable the older adult to have easy access to his or her LSB so that s/he can show to the significant others.
- d. Be sensitive to the older adult's response looking at his or her LSB, and be watchful for any negative moods or behaviours.
- e. Always empower the older adult to "own" his/her life story by asking permission to see the book.
- f. Possible applications:
  - Identify the components of the older adult's past that are still present, abilities that can be incorporated into the current day's caregiving approaches and programmes.
  - An appreciation of the older adult's life story can enable live-in migrant caregivers to deepen their acceptance of today's care challenges or difficulties
  - Use the LSB as a distraction when the older adult exhibit difficult behaviours that need refocusing or moods that may respond to positive input.
  - Use the book as a basis for assessment when determining approaches and care interventions, such as the selection of a meaningful activity, food and music preferences.

#### 8. Final product

Participating older adults will receive a personalized 12-page laminated memory album consisting of biographical information. Each  $10 \times 12$  inch page includes a 6-10 word declarative sentence printed in 60-70 size font for Chinese characters. Color or black and white photographs, drawings or newspaper cuttings illustrate the statement. The LSBs may contain personal pictures of their wedding and family, if older adults so desire.

Table 1. Standardized questions for LSB categories

| Ca | tegory | Standard questions | Remarks |
|---|---|---|---|
| 1. | Family, | Who else is in your family? | |
| | roots/ancestry | Where do you come from? Where is your home | |
| | | town? Is there any special product that comes | |
| | | from your home town? Any special place to see? | |
| | | Did you ever go back and visit? | |
| 2. | Religion | Do you practice ancestor worship? | |
| 3. | Childhood | Where did you live? | |
| | | Any interesting things to tell me about your | |
| | | childhood? | |
| | | What games did you play with your neighbors? | |
| | | Did you help your family at home? | |
| 4. | Education | Did you go to school? | |
| 5. | Marriage | Were you married? | If, prior to the sessions, |
| | | Did you choose a Western or a traditional | you already knew that |
| | | Chinese wedding? | the older adult is/was |
| | | | married, you can then ask |
| | | | him/her about his/her |
| | | | marriage. If the older |
| | | | adult has never been |
| | | | married, you may not |
| | | | need to ask (as some may |
| | | | find it offensive to be |
| | | | asked such a question). If |
| | | | the older adult never |
| | | | married because of |
| | | | special circumstances |
| | | | (e.g. the customs of a |
| | | | particular area), your |
| | | | approach and treatment |
| | | | of this topic can be |
| | | | dependent on the older |
| | | | adult's response in this |
| | | | area. |
| 6. | Place lived | When did you come to Hong Kong? | |
| | | Where did you live then? | |
| | | Which place did you live longest in making it your | |
| | | home? | |
| | | Any special features about the place you live? | |

| 7. | Close friends / | Were your neighbours/friends nice people? | |
|---|---|---|---|
| | neighbours | Did you go out together a lot? | |
| | | Did you watch out for each other? | |
| 8. | Work history | Did you work before? | The live-in migrant |
| | | What did you do for a living? | worker must be sensitive |
| | | Was the pay good? | to the response of the |
| | | | older adult, because most |
| | | | of our older adult have |
| | | | experienced hardships |
| | | | when they were young. If |
| | | | the level of income is |
| | | | especially meaningful to |
| | | | the older adult, e.g. s/he |
| | | | gave all his/her income to |
| | | | the family, then the live- |
| | | | in migrant caregivers can |
| | | | safely proceed. |
| 9. | Military history | Did you join the war or any wars? | |
| | | Were you a soldier? | |
| 10. | Awards | Did you win any award(s)? When? | |
| 11. | Lifestyle & | a. Interest and hobbies | |
| | hobbies | - What did you like to do most in the past? | |
| | | b. Travel | |
| | | <ul> <li>Did you ever go to visit other places?</li> </ul> | |
| | | c. Favorite foods & recipes | |
| | | - What is your favorite dishes? | |
| | | - What did you like to cook? | |
| | | d. Holidays/festivals/seasons of the year | |
| | | - What are some of the important festivals | |
| | | in a year? | |
| | | - Which one do you like best? | |
| | | - How to celebrate? | |
| | | - Did you do anything special on public | |
| | | holidays? | |
| | | - Which is your favorite season? | |
| | | e. Involvement in clubs and groups, position of | |
| | | leadership | |
| | | - For example, which church did you belong | |
| | | to? | |
| | | f. Volunteer experiences or community service | |

- Did you participate in any voluntary services?
- Whom did you serve?

#### g. Politics

- Did you take part in any political activity?
- For example, like joining the communist or the national party?
- h. Interest in literature and reading
  - What kind of literature do you like to read? Give examples, such as novels, poetry, prose.
  - Who is your favorite writer? Give examples, such as Li Bai, Du Fu, Bai Xian Yong, Jin Yong.
- i. Interest in music and creative arts
  - What kind of music do you like to listen to? Give examples, such as Chinese opera, classical music, pop songs.
  - What kinds of instruments do you play?
     Give examples, such as er hu.
  - What is your favorite art form? Give examples, such as engraving, calligraphy, water color painting.
- j. Animals and pets
  - What animals do you like as pets?
  - Did you have one?

### Protocol of training student helper/research assistant as the interpreter in the activities

Modified from Lai, C.K.Y. (2003). Improving the quality of life for nursing home residents with dementia: a life story approach. Dissertation: The University of Hong Kong.

1. The role of student helper/research assistant in the activities

There are an equal number of characters involved – an older adult, a live-in migrant caregivers, and a student helper/research assistant, in both the life storybook (LSB) intervention and control condition. For both activities, the older adult is the main character. The student helper/research assistant only plays a facilitative role in communication, by serving as an interpreter. It is because live-in migrant caregivers may not totally understand Cantonese which is the major dialect spoken by older adults in Hong Kong, and older adult may not understand English spoken by live-in migrant workers. In each of the activities, the live-in migrant caregiver will lead the activity and encourage the older adult to enjoy the social activity (for control group) or participate in the LSB production (for intervention group).

The student helper/research assistant is expected to assist in monitoring the compliance of the live-in migrant caregiver in delivering the activities using the checklist (Appendix VI).

- 2. Key points when working on the older adults and live-in migrant caregivers
  - a. Consider yourself as an integral member in the activity and be a friend to the older adult and the live-in migrant caregiver.
  - b. Avoid being overly active in taking part (e.g. instructing the older adult/live-in migrant caregiver to follow what you do).
  - c. Try to interpret the actual meaning of the sentences spoken by the older adult and live-in migrant caregiver without distorting the meaning.
- 3. Outline of training workshop for student helper/research assistant

| 2-hour workshop | Theme(s) |
|-----------------|-----------------------------------------------------------|
| First workshop | 1. Normal ageing |
| | 2. Introduction to mild cognitive impairment and dementia |
| | 3. Experience in caregiving older adults |
| Second workshop | 1. Introduction of the project |
| | 2. Communication skills with older adults |
| | 3. Compliance monitoring techniques |

# **Demographic & socioeconomic characteristics of the migrant carer**

| 1. Age | 2. Date of bir | th: day/ | month/ | year |
|---|---|---|---|---|
| 3. Sex ☐ Male ☐ Fer | male | | | |
| 4. Nationality | | | | |
| 5. Marital status | | | | |
| ☐ Single ☐ Married | ☐ Divorced | ☐ Widowed | | |
| 6. a) Education level | | | | |
| ☐ No schooling/ pre-prim | nary | nry | | |
| ☐ Secondary ☐ Terti | ary | | | |
| b) How many years of educ | cation do you ha | ve?Years | | |
| 7. a) Number of older peo | ple being cared | by you now | | |
| ☐ One | ☐ Two | □Three | ☐Four or more | |
| b) Living arrangement | | | | |
| ☐ live-out | | | | |
| ☐ live-in (Please go to o | question 7c) | | | |
| c) How many people are liv | ing with you in | the same apartm | ent? | |
| ☐ One | | | | |
| ☐ Two | | | | |
| ☐ Three | | | | |
| ☐ Four or more | | | | |
| 8. Caregiving experience | (inclusive all the | e past jobs) ? | | |
| Year(s)Month(s | ) | | | |
| 9. Caregiving experience | in Hong Kong ? | | | |
| Year(s)Month(s) | ı | | | |

# **Demographic and socioeconomic characteristics of the elderly**

| 1. Age | 2. Date of bi | rth : day/ | month/ | year | |
|---|---|---|---|---|---|
| 3. Sex ☐ Male ☐ Fe | male | | | | |
| 4. Nationality | | | | | |
| 5. Marital status | | | | | |
| ☐ Single ☐ Married | ☐ Divorced | ☐ Widowed | | | |
| 6. a) Education level | | | | | |
| ☐ No schooling/ pre-prin | nary | nary | | | |
| ☐ Secondary ☐ Tert | iary | | | | |
| b) How many years of educ | cation did the el | derly have? | Years | | |
| 7. Current living status | | | | | |
| a) Are you living alone? [ | ☐Yes (skip to q | uestion 6) \(\sigma\)No | | | |
| b) Who are you living with | now (select all | applicable)? | | | |
| i) 🗖 Living with spou | ise | ii) 🗖 Living with | child | iii) 🗖 Living with mai | d |
| iv) Living with oth | er people who | are not spouse or cl | hild | | |
| ( Please specify the re | elationship of th | ose people with eld | derly) | | |
| c) Type of Housing | | | | | |
| ☐ Rent public hou | sing $\square$ | Self-owned public | housing | ☐ Rent private housing | |
| ☐ Self-owned priv | ate housing | ☐ Old age h | ome | | |
| ☐ Others (please s | pecify: | ) | | | |

| 8. a) Employment | | | | |
|---|---|---|---|---|
| ☐ Unemployed | ☐ Retire | d | | |
| ☐ Employed | | | | |
| ☐ Full Time | | | | |
| ☐ Part time | | | | |
| ☐ Temporary | | | | |
| b) Occupation (Past/Curr | rent) | | | |
| ☐ Managers and administr | rators | ☐ Professionals | | ☐ Associate professionals |
| ☐ Clerical support worker | S | ☐ Service and sales worker | rs | ☐ Craft and related workers |
| ☐ Plant and machine opera | ators and | ☐ Elementary occupations | | ☐ Others (Please specify: |
| assemblers | | | | ) |
| 9. Have the elderly been dia | agnosed by m | edical doctor with the follow | ing disea | ase(s)? |
| ☐ Hypertension | ☐ Diabetes | | □ Нур | erlipidemia |
| ☐ Heart disease | ☐ Osteopor | osis | ☐ Arth | ritis |
| ☐ Parkinson's Disease | ☐ Asthma | | ☐ Can | cer |
| | | | (Please | specify) |
| ☐ Depression | ☐ Mental il | lness other than depression | ☐ Othe | ers |
| □Dementia | (Please spec | ify) | (Please | specify) |
| (Mild / Moderate/ Late) | | | | |

# **Focus group interview**

| The inte | erview may follow the questions: |
|---|---|
| 1. | Would you please tell me your experiences/opinions with regard to learning and participating in the intervention? |
| 2. | Would you please tell whether participating in the intervention has made a difference or not in relation to your relationship with the live-in migrant care worker/older adult? |
| 3. | What were the challenges in conducting LSB with older adults? How did you solve those challenges |
| 4. | Any other comments/suggestions based on your participation in the intervention? |

# **Checklist for monitoring the intervention fidelity**

Modified from Lai, C.K.Y. (2003). Improving the quality of life for nursing home residents with dementia: a life story approach. Dissertation: The University of Hong Kong.

LSB intervention / Social activities\* (delete as appropriate)

| Name of reviewer: | |
|---|---|
| Name of the live-in migrant worker being reviewed: | |
| Date of review: | (1 <sup>st</sup> /2 <sup>nd</sup> /3 <sup>rd</sup> /4 <sup>th</sup> session*) |

Please tick "V" whether the live-in migrant caregiver achieve the item listed in the table.

| | | Yes | No |
|---|---|---|---|
| | Preparing the session | | |
| | Sufficient planning for what to do in the session | | |
| | Preparation beforehand, e.g. has appropriate pictures ready, not saying that she | | |
| | forgot to do this or that, etc. | | |
| Structure | Not over-doing things for the older adult, not having to make the older adult wait or | | |
| Struc | showing indecision | | |
| | Usage of material | | |
| | A wide variety of material used (pictures, news clippings, photos) | | |
| | Use of words (tendency to use more words or more pictures) | | |
| | Use of appropriate pictures | | |
| | General attitude | | |
| | Facilitative | | |
| | Encouraging | | |
| | Directive but not domineering | | |
| | Communication | | |
| | Behaviours | | |
| | - Smiles | | |
| Process | - Uses appropriate body language, e.g. leans toward older adult | | |
| Pro | - Positive regard for older adult and interpreter | | |
| | - Non-judgmental attitude toward older adult behavior | | |
| | - Sensitive to needs of older adult | | |
| | Skills used | | |
| | - Positive reinforcement | | |
| | - Active listening | | |
| | - Paraphrasing | | |
| | - Use of open-ended questions | | |

| | - Closed-ended questions used appropriately |
|---|---|
| | Processes skills |
| | Time control |
| | Has three stages in process: |
| | - Introduction (summary of previous session, introducing this session) |
| | - Body (tasks for today) |
| | - Closure (summary of what have been done today and what will come in the |
| | next sessions) |
| | Involvement of the older adult |
| | Allows time for expression |
| | Provides opportunities for involvement, e.g. cutting of pictures, arranging pictures; |
| | allows older adult to choose |
| | Ensure that older adult is using the necessary aids, e.g. hearing aid, spectacles, or |
| | magnifying glasses |
| Outcome | Reference to protocol |
| | Adherence to protocols |
| | Reference to categories of LSB – lifestyle and life course approach |
| | End product |
| | LSB categories by and large the same |
| | Choice of words, use of pictures by and large similar |
| | Font size and color used by and large alike |